CLINICAL TRIAL: NCT02246062
Title: Impact of Preanesthetic Information and Behavioral Intervention Using Smartphone Application on Anxiety of Children
Brief Title: Impact of Preanesthetic Information and Behavioral Intervention Using Smartphone on Anxiety of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Débora de Oliveira Cumino, MSC, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 288.712
Record Dates: First submitted 2014-03-20; First posted 2014-09-22 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Anxiety State; Parent-Child Relations
Keywords: Anxiety; Anesthesia; Evaluation; Preoperative care; Child
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (No Intervention): in which the relative receive only conventional verbal information one day before the procedure at ward.
- info group (Active Comparator): in which the relative, in addition to conventional verbal information, received a leaflet containing information about the anesthetic procedure one day before the surgery at ward.
  Interventions: Behavioral: info
- smartphone group (Active Comparator): in which the relative received only conventional verbal information one day before the procedure and the child received smartphone application immediately before entering the operating room
  Interventions: Behavioral: smartphone
- smartphone and info group (Active Comparator): in which the relative, in addition to conventional verbal information, received a leaflet containing information about the anesthetic procedure one day before the surgery and the child received smartphone application immediately before entering the operating room.
  Interventions: Behavioral: info; Behavioral: smartphone

INTERVENTIONS:
Behavioral: info — the relative received leaflet containing information about the anesthetic procedure one day before the surgery at ward.
  Arms: info group; smartphone and info group
Behavioral: smartphone — the child received smartphone application immediately before entering the operating room
  Arms: smartphone and info group; smartphone group

SUMMARY:
Background: Preoperative Anxiety is a negative factor in anesthetic and surgical experience. Among the strategies for reducing children's anxiety, non-pharmacological strategies are as important as the pharmacological ones, but their its validity is still controversial.

Objectives: The aim of this study is to verify if the information provided to relatives as well as and smartphone application provided to children interferes in prevalence and level of child preoperative anxiety.

Methods: Eighty four children, 4-8 years old, ASA I, II and III, undergoing elective surgical procedures and their relatives are randomly allocated into four groups: control group (CG) where the relative received conventional information about anesthesia; info group (IG), relative received an information leaflet about anesthesia; device group (DG), relative received only conventional verbal information and the child received smartphone application immediately before entering the operating room; device and info group (DIG) relative received a leaflet containing information and the child received smartphone application. Children's anxiety will be assessed using the modified Yale Preoperative Anxiety Scale (m-YPAS) on three occasions: at the ward (W), surgical theater in the waiting room (WR) and at the operating room (OR). Statistics analysis will employ by Kruskall-Wallis and Mann-Whitney tests for prevalence and level of anxiety in the groups.

DETAILED DESCRIPTION:
Introduction

Intense preoperative anxiety in children has been associated with difficulty in anesthetic induction. In addition, anxiety of relatives is a factor of great importance and influence on the preoperative anxiety levels of children and effectively contributes to the development of behavioral changes in postoperative period.

Distress before surgery has been associated with short- and long-term consequences, including risks of emergence delirium and maladaptive postoperative behaviors. Strategies to decrease children's anxiety can provide suitable induction and minimizes these risks.

It is estimated that 40% to 75% of children undergoing surgery experience significant fear and anxiety during the preoperative period3-5 Several authors suggest that children under 4 years of age are at greater risk for developing anxiety preoperatively.

Among the strategies for reducing the pediatric population anxiety, the non-pharmacological approaches through alternative therapies that act on the psychological aspects are as important as the pharmacological ones 9.

Currently, there is great motivation towards non-pharmacological interventions aimed at anxiety relief for children and their families, such as parental presence during induction of anesthesia (PPIA), educational programs to prepare the family, and written information on anesthetic procedure provided to relatives and/or children. This is due in part to the large growth in outpatient practice and increased participation and presence of parents during children's hospitalization, but also to the new institutional strategies that motivate a more humane medical practice. Furthermore, there have emerged efficient behavioral intervention programs that use toys, cartoons, video games and smartphones.

It has been suggested the intuitive and easeness of use, and popularity, of smartphones as a way to make children become absorbed by scrolling through its menus, playing and investigating its other functions, hence making the anesthesiologists' approach trouble-free.

Some authors showed that using smartphone application and other electronic devices as part of a behavioral intervention program for children, while taking into account individual characteristics, may be a simple and effective way to reduce preoperative anxiety.

Objectives The aim of this study is to determine whether the quality of information provided to relatives at the ward and playing with age appropriate smartphone application may have an impact on prevalence and level of child's anxiety in the operating room (OR) at the induction of anesthesia.

Method

After approval by the Research Ethics Committee of Irmandade da Santa Casa de São Paulo, an open randomized clinical trial should be conducted to compare the level of anxiety of children and their relatives, according to the quality of information and use or not of smartphone application received in the preanesthetic period.

Eighty-four children undergoing elective surgical procedures and their relatives will be randomly selected through the List Randomizer program (www.random.org) and allocated into four groups: control group (CG), in which the relative receive only conventional verbal information one day before the procedure at ward; informative group (IG), in which the relative, in addition to conventional verbal information, received a leaflet containing information about the anesthetic procedure one day before the surgery at ward; smartphone group (SG), in which the relative received only conventional verbal information one day before the procedure and the child received smartphone application immediately before entering the operating room; smartphone and informative group (SIG) in which the relative, in addition to conventional verbal information, received a leaflet containing information about the anesthetic procedure one day before the surgery and the child received smartphone application immediately before entering the operating room.

Developed by the author, the leaflet consists of 17 brief items, such as questions and answers, and provides information regarding the most frequently asked questions by the relatives, as observed in our clinical practice. The contents of this informative leaflet cover aspects of the specialty and practice of anesthesiology, such as suspension and use of medications, fasting, full stomach and refeeding after anesthesia, laboratory tests, anesthesia in children, types of anesthesia, risks, induction and recovery room, presence of parents, and how to contribute to a peaceful anesthesia in children.

Inclusion criteria are ASA physical status I, II and III, according to the classification of the American Society of Anesthesiologists (ASA), age between 4 and 8 years, undergoing minor-medium elective surgical procedures with an indication of general anesthesia, who shall not receive premedication and whose parents are not illiterate.

The exclusion criteria for children are psychomotor deficits, use of psychoactive drugs, hearing and visual impairment, previous surgery; and for relatives, the exclusion criteria are illness or mental disorder clinically recognized and decline to participate.

The study begins always in the ward (W), one day before the procedure, during preanesthesia evaluation and on the conventional provision of information about anesthesia. One of the researchers applies the observational m-YPAS scale for child and then the relatives are fully informed about the characteristic of the study and will be asked to sign the consent form. At the end of the preanesthetic evaluation (APA) the relatives of the IG and SIG groups receive an information leaflet.

At the day of the procedure, in the waiting room (WR) of surgical centers, before the child is taken to the operating room (OR), the child anxiety is assessed by m-YPAS scale. All groups will also answer a sociodemographic questionnaire and open statement for satisfaction about the information received. The children of the groups SG and SIG, before taken to the OR receive smartphones for playing, remaining always accompanied by the relatives until the end of induction. In the OR, all children undergo standard monitoring and, immediately before induction of anesthesia through conventional technique (either intravenous or inhalational), are re-evaluated using m-YPAS (OR time).

Level and prevalence of children's anxiety (m-YPAS), will be measured at three times: ward (W), waiting room (WR) and operating room (OR) immediately before induction. The observational m-YPAS was used as originally proposed by Kain et al. A partial score was given for each domain, based on the score observed by the researcher, divided by the number of categories in that domain. The score for each domain is added to the others and then multiplied by 20. Cut-off scores to classify patients are: without anxiety (23.4-30), with anxiety (< 30).

For sample size calculation, it was considered that the prevalence of children's anxiety in the operating room is 75% 23 and that the proposed intervention is able to reduce it by 35% 15. Thus, the investigators propose to use α-error of 5%, β-error of 20%, and confidence interval of 95%, totaling 84 patients, 21 in each group.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II and III a
* age between 4 and 8 years
* undergoing minor-medium elective surgical procedures
* indication of general anesthesia
* not receive premedication
* parents are not illiterate.

Exclusion Criteria:

* psychomotor deficits
* use of psychoactive drugs
* hearing and visual impairment
* previous surgery
* for relatives, illness or mental disorder clinically recognized and decline to participate.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ligia AS Mathias, PhD, Study Director — Irmandade Santa Casa de Misericórdia de São Paulo
Locations (1):
- Irmandade Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Melamed BG, Siegel LJ. Reduction of anxiety in children facing hospitalization and surgery by use of filmed modeling. J Consult Clin Psychol. 1975 Aug;43(4):511-21. doi: 10.1037/h0076896. No abstract available. PMID 1159149
- [Background] Lumley MA, Melamed BG, Abeles LA. Predicting children's presurgical anxiety and subsequent behavior changes. J Pediatr Psychol. 1993 Aug;18(4):481-97. doi: 10.1093/jpepsy/18.4.481. PMID 8410571
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] ECKENHOFF JE. Relationship of anesthesia to postoperative personality changes in children. AMA Am J Dis Child. 1953 Nov;86(5):587-91. doi: 10.1001/archpedi.1953.02050080600004. No abstract available. PMID 13103772
- [Background] Watson AT, Visram A. Children's preoperative anxiety and postoperative behaviour. Paediatr Anaesth. 2003 Mar;13(3):188-204. doi: 10.1046/j.1460-9592.2003.00848.x. No abstract available. PMID 12641680
- [Background] Bevan JC, Johnston C, Haig MJ, Tousignant G, Lucy S, Kirnon V, Assimes IK, Carranza R. Preoperative parental anxiety predicts behavioural and emotional responses to induction of anaesthesia in children. Can J Anaesth. 1990 Mar;37(2):177-82. doi: 10.1007/BF03005466. PMID 2311148
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Kain ZN, Mayes LC, Weisman SJ, Hofstadter MB. Social adaptability, cognitive abilities, and other predictors for children's reactions to surgery. J Clin Anesth. 2000 Nov;12(7):549-54. doi: 10.1016/s0952-8180(00)00214-2. PMID 11137417
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Saadat H, McClain B, Wang SM. Predicting which children benefit most from parental presence during induction of anesthesia. Paediatr Anaesth. 2006 Jun;16(6):627-34. doi: 10.1111/j.1460-9592.2006.01843.x. PMID 16719878
- [Background] Kain ZN, Caldwell-Andrews AA, Mayes LC, Weinberg ME, Wang SM, MacLaren JE, Blount RL. Family-centered preparation for surgery improves perioperative outcomes in children: a randomized controlled trial. Anesthesiology. 2007 Jan;106(1):65-74. doi: 10.1097/00000542-200701000-00013. PMID 17197846
- [Background] Astuto M, Rosano G, Rizzo G, Disma N, Raciti L, Sciuto O. Preoperative parental information and parents' presence at induction of anaesthesia. Minerva Anestesiol. 2006 Jun;72(6):461-5. PMID 16682916
- [Background] Wright KD, Stewart SH, Finley GA, Buffett-Jerrott SE. Prevention and intervention strategies to alleviate preoperative anxiety in children: a critical review. Behav Modif. 2007 Jan;31(1):52-79. doi: 10.1177/0145445506295055. PMID 17179531
- [Background] Chundamala J, Wright JG, Kemp SM. An evidence-based review of parental presence during anesthesia induction and parent/child anxiety. Can J Anaesth. 2009 Jan;56(1):57-70. doi: 10.1007/s12630-008-9008-3. Epub 2008 Dec 20. PMID 19247779
- [Background] Lee J, Lee J, Lim H, Son JS, Lee JR, Kim DC, Ko S. Cartoon distraction alleviates anxiety in children during induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1168-73. doi: 10.1213/ANE.0b013e31824fb469. Epub 2012 Sep 25. PMID 23011563
- [Background] Mifflin KA, Hackmann T, Chorney JM. Streamed video clips to reduce anxiety in children during inhaled induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1162-7. doi: 10.1213/ANE.0b013e31824d5224. Epub 2012 Oct 9. PMID 23051880
- [Background] Lee JH, Jung HK, Lee GG, Kim HY, Park SG, Woo SC. Effect of behavioral intervention using smartphone application for preoperative anxiety in pediatric patients. Korean J Anesthesiol. 2013 Dec;65(6):508-18. doi: 10.4097/kjae.2013.65.6.508. Epub 2013 Dec 26. PMID 24427456
- [Background] Low DK, Pittaway AP. The 'iPhone' induction - a novel use for the Apple iPhone. Paediatr Anaesth. 2008 Jun;18(6):573-4. doi: 10.1111/j.1460-9592.2008.02498.x. Epub 2008 Feb 28. No abstract available. PMID 18312515
- [Background] Kerimoglu B, Neuman A, Paul J, Stefanov DG, Twersky R. Anesthesia induction using video glasses as a distraction tool for the management of preoperative anxiety in children. Anesth Analg. 2013 Dec;117(6):1373-9. doi: 10.1213/ANE.0b013e3182a8c18f. PMID 24257388
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Marcolino JA, Mathias LA, Piccinini Filho L, Guaratini AA, Suzuki FM, Alli LA. Hospital Anxiety and Depression Scale: a study on the validation of the criteria and reliability on preoperative patients. Rev Bras Anestesiol. 2007 Feb;57(1):52-62. doi: 10.1590/s0034-70942007000100006. English, Portuguese. PMID 19468618
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Cumino Dde O, Cagno G, Goncalves VF, Wajman DS, Mathias LA. Impact of preanesthetic information on anxiety of parents and children. Braz J Anesthesiol. 2013 Nov-Dec;63(6):473-82. doi: 10.1016/j.bjane.2013.04.003. Epub 2013 Dec 5. PMID 24565345
- [Derived] Cumino DO, Vieira JE, Lima LC, Stievano LP, Silva RA, Mathias LA. Smartphone-based behavioural intervention alleviates children's anxiety during anaesthesia induction: A randomised controlled trial. Eur J Anaesthesiol. 2017 Mar;34(3):169-175. doi: 10.1097/EJA.0000000000000589. PMID 28146459

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Info Group | Smartphone Group | Smartphone and Info Group
Started | 21 | 21 | 21 | 21
Completed | 21 | 21 | 21 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Info Group | Smartphone Group | Smartphone and Info Group | Total
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.29 (1.15) | 5.45 (1.0) | 5.29 (0.96) | 5.65 (1.04) | 5.41 (1.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 7 | 2 | 25
  Male | 14 | 12 | 14 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Impact of Preanesthetic Information and Behavioral Intervention Using Smartphone Application on Anxiety of Children Measure by m-YPAS.
Description: The level of child's anxiety will be measure by modified Yale Preoperative Anxiety Scale (m-YPAS). The total score of m-YPAS was calculated according to what was originally proposed by Kain et al. The total scores range from 23,4 until 100. Cut-off scores to classify patients with or without anxiety were: without anxiety (23.4 - 30), with anxiety (< 30).
Time Frame: 24 hours before surgery
Measure: Mean (Standard Deviation); unit: units on a scale m-YPAS
Arm/Group | Control Group | Info Group | Smartphone Group | Smartphone and Info Group
Number analyzed (Participants) | 21 | 21 | 21 | 21
units on a scale m-YPAS | 27.8 (10.26) | 24.18 (2.12) | 23.79 (1.27) | 24.98 (6.20)

2. Other Pre Specified Outcome: Impact of Preanesthetic Information and Behavioral Intervention Using Smartphone Application on Anxiety of Children Measure m-YPAS.
Description: The level of child's anxiety will be measure by modified Yale Preoperative Anxiety Scale (m-YPAS). The total score of m-YPAS was calculated according to what was originally proposed by Kain et al. The total scores range from 23,4 until 100. Cut-off scores to classify patients with or without anxiety were: without anxiety (23.4 - 30), with anxiety (> 30).
Time Frame: Immediately before entering operation room
Measure: Mean (Standard Deviation); unit: units on a scale m-YPAS
Arm/Group | Control Group | Info Group | Smartphone Group | Smartphone and Info Group
Number analyzed (Participants) | 21 | 21 | 21 | 21
units on a scale m-YPAS | 31.88 (13.94) | 23.88 (2.18) | 25.85 (6.44) | 25.93 (9.05)

3. Other Pre Specified Outcome: Impact of Preanesthetic Information and Behavioral Intervention Using Smartphone Application on Anxiety of Children Measure by m-YPAS.
Description: as for outcome 2
Time Frame: Immediately before induction of anesthesia
Measure: Mean (Standard Deviation); unit: units on a scale m-YPAS
Arm/Group | Control Group | Info Group | Smartphone Group | Smartphone and Info Group
Number analyzed (Participants) | 21 | 21 | 21 | 21
units on a scale m-YPAS | 51.13 (23.65) | 30.29 (14.40) | 36.55 (19.08) | 28.23 (10.47)

ADVERSE EVENTS:
Time Frame: 1 day
Description: adverse event assessment was based on drop out rate
Arm/Group | Control Group | Info Group | Smartphone Group | Smartphone and Info Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No